CLINICAL TRIAL: NCT00948337
Title: A Randomized Controlled Trial on the Effect of Intervention With Health Educational Material on Knowledge, Attitude, and Behavior in Cancer Survivors
Brief Title: A Study With Health Educational Material on Health Promotion in Cancer Survivors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: National Cancer Center, National Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NCS-09-266
Record Dates: First submitted 2009-07-28; First posted 2009-07-29 (Estimated); Last update posted 2010-02-26 (Estimated); Status verified 2009-09

CONDITIONS: Stomach Cancer; Colon Cancer; Thyroid Cancer; Breast Cancer
MeSH Terms: conditions — Stomach Neoplasms; Colonic Neoplasms; Thyroid Neoplasms; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Photonovella of Secondary Cancer Screening (Experimental)
  Interventions: Behavioral: Brochure of Secondary Cancer Screening
- Photonovella of Dietary Suppelment of Cancer survivor (Active Comparator)
  Interventions: Behavioral: Brochure of Secondary Cancer Screening

INTERVENTIONS:
Behavioral: Brochure of Secondary Cancer Screening — One kind of printed educational material

SUMMARY:
The purpose of this study is to provide educational material to promote screening for second primary cancer for the intervention group, or educational material to instruct appropriate use of dietary supplement for the control group.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18, <80
* Cancer survivors (pathologically confirmed)
* Finished primary treatment (surgery, radiotherapy, chemotherapy)
* >= 1 year from cancer diagnosis
* No evidence of recurrence, metastasis, and second primary cancer
* No evidence of hereditary cancer
* ECOG 0,1,2
* Ability in reading Korean educational material

Exclusion Criteria:

* ECOG 3,4
* Disagree with the investigators study purpose

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Estimated)
Dates: Start 2009-08; Primary Completion 2009-11 (Actual); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Screening behavior for second primary cancer | After 1 yr

SECONDARY OUTCOMES:
Knowledge and attitudes of Secondary cancer screening and dietary supplement | In 2 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Samsung Medical Center, Seoul

REFERENCES:
- [Derived] Shin DW, Cho J, Kim YW, Oh JH, Kim SW, Chung KW, Lee WY, Lee JE, Guallar E, Lee WC. Efficacy of an educational material on second primary cancer screening practice for cancer survivors: a randomized controlled trial. PLoS One. 2012;7(3):e33238. doi: 10.1371/journal.pone.0033238. Epub 2012 Mar 29. PMID 22479375